CLINICAL TRIAL: NCT03436862
Title: A Phase II Single Arm Study of Nivolumab as Maintenance Therapy After Autologous Stem Cell Transplantation in Patients With Hodgkin Lymphoma at Risk of Relapse or Progression
Brief Title: Nivolumab Maintenance Therapy After Autologous Stem Cell Transplant in Hodgkin Lymphoma Pts at Relapse/Progression Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BMT 24
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-06

CONDITIONS: Hodgkin Lymphoma
Keywords: Nivolumab; Autologous Stem Cell Transplant; Blood cancers
MeSH Terms: conditions — Hodgkin Disease; Hematologic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Patients will receive Nivolumab 240 mg by intravenous infusion (IV) starting Day 45-120 post-transplant (±10 days) every 2 weeks for up to a maximum of 6 months of treatment.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 240 mg IV infusion over 60 minutes given every 2 weeks for up to 6 months.
  Other Names: Opdivo

SUMMARY:
This is a Phase II single-arm open-label study of nivolumab as maintenance therapy after autologous stem cell transplantation in patients with Hodgkin lymphoma at risk of relapse or progression.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate safety and tolerability of nivolumab as maintenance therapy early after autologous stem cell transplant in patients with Hodgkin's Lymphoma (HL).

Eligible patients will receive nivolumab (240 mg IV) every 2 weeks (± 2 days as long as interval between doses is 12-16 days) starting 45-120 post-transplant for up to a maximum of 6 months of treatment. Response to treatment will be assessed 6 months and 1 year post-transplant using Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older with Hodgkin Lymphoma who have received auto-HSCT in the previous 45-120 days.
* Complete response (CR), partial response (PR) or stable disease (SD) to salvage therapy prior to ASCT.
* High risk of residual HL post-ASCT, as determined by 1 of the following:

  * Positive positron emission tomography (PET) scan defined by the Deauville scale 3-4 and within 2 months of start of high dose chemotherapy prior to ASCT
  * Refractory to frontline therapy
  * Relapse <12 months after frontline therapy
  * Relapse ≥12 months after frontline therapy with extra-nodal disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 - 1.
* Adequate hematologic function defined as all of the following:

  * Absolute neutrophil count (ANC) ≥1000/μL
  * Hemoglobin (Hgb) ≥8 g/dL (transfusions to reach this point are not permitted)
  * Platelets ≥50,000/μL (transfusion is not permitted)
* Adequate liver function defined as all of the following:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN)
  * Total bilirubin ≤1.5 x ULN (unless the patient has Grade 1 bilirubin elevation due to Gilbert's disease or a similar syndrome involving slow conjugation of bilirubin)
* Adequate renal function defined as serum creatinine ≤1.5 mg/dL (133 μmol/L).
* Females of childbearing potential must have a negative serum or urine pregnancy test result within 72 hours prior to the first dose of nivolumab and must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab and for 7 months following their last dose of study drug. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.
* Male patients with female partners of childbearing potential and women patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 7 months following last dose of study drug. Male patients must also refrain from donating sperm during their participation in the study and for 7 months following last dose of study drug.

Exclusion Criteria:

* Patients that have received an allogenic transplant.
* Post-ASCT or current therapy with other anti-neoplastic or investigational agents.
* Best clinical response of progressive disease prior to ASCT.
* Patients with any autoimmune disease or a history of autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Use of a study drug ≤ 21 days or 5 half-lives (whichever is shorter) prior to the first dose of nivolumab. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of nivolumab is required.
* Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
* Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
* Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks prior to study entry and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
* Pregnant or lactating
* Acute or chronic liver, renal, or pancreatic disease.
* Uncontrolled diabetes mellitus. Patients with Type II diabetes are eligible if they require only oral hypoglycemic agents.
* Any of the following cardiac diseases currently or within the last 6 months:

  * Left Ventricular Ejection Fraction (LVEF) <45% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc interval >480 ms on screening electrocardiogram (ECG)
  * Unstable angina pectoris
  * Congestive heart failure (New York Heart Association (NYHA) ≥ Grade 2
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate- controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
  * Valvular disease with significant compromise in cardiac function
* Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] >180 mmHg or diastolic blood pressure (DBP) >100 mmHg) (patients with values above these levels must have their blood pressure (BP) controlled with medication prior to starting treatment).
* Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C. Testing at baseline is not required.
* Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bachier, MD, Study Chair — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - HCA Midwest, Kansas City, Missouri
  - Tennessee Oncology, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nivolumab
Started | 37
Completed | 31
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nivolumab
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 36 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events as a Measure of Safety and Tolerability of Nivolumab as Maintenance Therapy
Description: Adverse events will be graded according to National Cancer Institute Common Technology Criteria for Adverse Events (NCI CTCAE version 4.03).
Time Frame: Every 2 weeks up to a maximum of 6 months of treatment, then up to 100 days after treatment discontinuation
Population: All participants who have received at least one dose of study drug (Nivolumab) treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 37
Participants | 33

2. Secondary Outcome: Progression-free Survival (PFS) Kaplan-Meier Estimate at 12 Month Interval
Description: Kaplan-Meier PFS estimate at 12 month interval when nivolumab is administered as maintenance therapy. Progression-Free Survival (PFS), defined as the time from the first day of study drug administration (Day 1) to disease progression as defined by the Recommendations for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma: The Lugano Classification (Cheson et al. 2014), or death on study. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment.
Time Frame: 1 year after date of first dose of study drug for each patient
Population: All participants who have received at least one dose of study treatment (Nivolumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nivolumab
Number analyzed (Participants) | 37
percentage of participants | NA [NA to NA] — Since so few patients progressed or died, the median progression-free survival estimate at 12 months after first dose was not estimable by Kaplan-Meier method nor the 95% confidence interval.

ADVERSE EVENTS:
Time Frame: Serious and/or other adverse events were assessed from the date of first dose to 100 days after last dose of study treatment, up to approximately 280 days. All-Cause Mortality was monitored from date of consent to 2 years after last dose of study treatment, approximately 2.5 years.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03.
Arm/Group | Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/37
Serious Adverse Events (participants affected / at risk) | 4/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=37)
Pyrexia (General disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab (N=37)
Anaemia (Blood and lymphatic system disorders) | 4
Vertigo (Ear and labyrinth disorders) | 2
Vision blurred (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Catheter site pain (General disorders) | 2
Fatigue (General disorders) | 10
Pain (General disorders) | 3
Pyrexia (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Lymphocyte count decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03436862/Prot_SAP_000.pdf